CLINICAL TRIAL: NCT01185301
Title: A Double-Blind, Randomized, Parallel-Arm, Multicenter Study to Determine the Dose Response of Methotrexate (MTX) in Combination Therapy With Adalimumab in Subjects With Early Rheumatoid Arthritis (CONCERTO)
Brief Title: Study to Determine the Effects of Different Doses of Methotrexate (MTX) When Taken With Adalimumab in Subjects With Early Rheumatoid Arthritis (RA)
Acronym: CONCERTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-073; 2010-019514-24 (EudraCT Number)
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-09

CONDITIONS: Early Rheumatoid Arthritis
Keywords: Arthritis; Erosion; Humira; Adalimumab; Injection; Rheumatoid; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ADA + 2.5 mg MTX (Active Comparator): 2.5 mg methotrexate (MTX) oral capsule weekly with 40 mg adalimumab (ADA) subcutaneous (SC) injection every other week (EOW) for 26 weeks
  Interventions: Biological: adalimumab; Drug: methotrexate
- ADA + 5 mg MTX (Active Comparator): 5 mg MTX oral capsule weekly with 40 mg ADA SC injection EOW for 26 weeks
  Interventions: Biological: adalimumab; Drug: methotrexate
- ADA + 10 mg MTX (Active Comparator): 10 mg MTX oral capsule weekly with 40 mg ADA SC injection EOW for 26 weeks
  Interventions: Biological: adalimumab; Drug: methotrexate
- ADA + 20 mg MTX (Active Comparator): MTX oral capsule dose escalation from 10 mg to 20 mg in 2.5 mg increments every other week (10 mg x 2 weeks, 12.5 mg x 2 weeks, 15 mg x 2 weeks, 17.5 mg x 2 weeks), then 20 mg for 18 weeks with 40 mg ADA SC injection EOW for 26 weeks
  Interventions: Biological: adalimumab; Drug: methotrexate

INTERVENTIONS:
Biological: adalimumab — Pre-filled syringe every other week
  Other Names: Humira
Drug: methotrexate — weekly oral capsule dosing

SUMMARY:
The purpose of this study is to determine the effects of different doses of methotrexate (MTX) when taken with adalimumab in subjects with early rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age
* Subject has a diagnosis of Rheumatoid Arthritis (RA) as defined by either the 1987-revised American College of Rheumatology (ACR) classification criteria or the new ACR/ European League Against Rheumatism (EULAR) diagnostic criteria for RA 2010 and has a disease duration of less than 1 year from diagnosis by a licensed health care provider
* Subject must meet the following criteria:

  1. Disease Activity Score of C-reactive Protein (DAS28[CRP]) ≥ 3.2 (at the Baseline visit only)
  2. At least 6 swollen joints out of 66 assessed (at the Screening and Baseline visits)
  3. At least 8 tender joints out of 68 assessed (at the Screening and Baseline visits)
  4. C-reactive protein (CRP) ≥ 1.5 mg/dL (at the Screening visit only), or erythrocyte sedimentation rate (ESR) ≥ 28 mm/1h (at the Screening and Baseline visits)
  5. Fulfill at least one of the following three criteria: Rheumatoid Factor (RF) positive, have at least 1 bony erosion, anti-cyclic citrullinated peptide (anti-CCP) antibody positive
* Subject is judged to be in good health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, physical examination, chest x-ray (CXR), and a 12-lead electrocardiogram (ECG) performed during Screening

Exclusion Criteria:

* Subject has previous exposure to any systemic biologic therapy including adalimumab
* Subject has been previously treated with greater than 1 disease modifying antirheumatic drugs (DMARDs) or with methotrexate (MTX)
* Subject has undergone joint surgery within the preceding two months (at joints to be assessed within the study)
* Subject has chronic arthritis diagnosed before age 17 years
* History of invasive infection (e.g., listeriosis and histoplasmosis), chronic or active Hepatitis C infection, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active tuberculosis (TB)
* Hepatitis B virus: hepatitis B surface antigen (HBs Ag) positive (+) or detected sensitivity on the hepatitis B virus DNA (HBV DNA) polymerase chain reaction (PCR) qualitative test
* Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the Baseline Visit or oral anti-infectives within 14 days prior to the Baseline visit
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Carlson, MD, Study Director — AbbVie
Locations (68):
- United States (30):
  - Site Reference ID/Investigator# 38973, Huntsville, Alabama
  - Site Reference ID/Investigator# 41962, Mesa, Arizona
  - Site Reference ID/Investigator# 39260, Phoenix, Arizona
  - Site Reference ID/Investigator# 45323, Little Rock, Arkansas
  - Site Reference ID/Investigator# 38912, Hemet, California
  - Site Reference ID/Investigator# 39673, Victorville, California
  - Site Reference ID/Investigator# 38909, Jacksonville, Florida
  - Site Reference ID/Investigator# 40422, Miami, Florida
  - Site Reference ID/Investigator# 38910, Sarasota, Florida
  - Site Reference ID/Investigator# 44284, Atlanta, Georgia
  - Site Reference ID/Investigator# 38907, Gainesville, Georgia
  - Site Reference ID/Investigator# 38972, Lawrenceville, Georgia
  - Site Reference ID/Investigator# 39670, Rock Island, Illinois
  - Site Reference ID/Investigator# 42282, Springfield, Illinois
  - Site Reference ID/Investigator# 38911, Wichita, Kansas
  - Site Reference ID/Investigator# 39672, Covington, Louisiana
  - Site Reference ID/Investigator# 42204, Omaha, Nebraska
  - Site Reference ID/Investigator# 40651, Clifton, New Jersey
  - Site Reference ID/Investigator# 41422, Freehold, New Jersey
  - Site Reference ID/Investigator# 41424, The Bronx, New York
  - Site Reference ID/Investigator# 40463, Greenville, North Carolina
  - Site Reference ID/Investigator# 42202, Columbus, Ohio
  - Site Reference ID/Investigator# 44282, Norman, Oklahoma
  - Site Reference ID/Investigator# 41423, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 38971, Charleston, South Carolina
  - Site Reference ID/Investigator# 39666, Jackson, Tennessee
  - Site Reference ID/Investigator# 39643, Dallas, Texas
  - Site Reference ID/Investigator# 45325, Dallas, Texas
  - Site Reference ID/Investigator# 52042, Houston, Texas
  - Site Reference ID/Investigator# 40602, Seattle, Washington
- Argentina (4):
  - Site Reference ID/Investigator# 44924, Buenos Aires
  - Site Reference ID/Investigator# 44926, Buenos Aires
  - Site Reference ID/Investigator# 44925, Rosario, Santa Fe
  - Site Reference ID/Investigator# 47302, San Juan
- Austria (3):
  - Site Reference ID/Investigator# 44928, Graz
  - Site Reference ID/Investigator# 44930, Vienna
  - Site Reference ID/Investigator# 44927, Vienna
- Belgium (4):
  - Site Reference ID/Investigator# 44934, Brussels
  - Site Reference ID/Investigator# 44935, Genk
  - Site Reference ID/Investigator# 44933, Gilly
  - Site Reference ID/Investigator# 44932, Liège
- Canada (2):
  - Site Reference ID/Investigator# 43783, Edmonton
  - Site Reference ID/Investigator# 43782, Winnipeg
- Czechia (6):
  - Site Reference ID/Investigator# 44937, Brno
  - Site Reference ID/Investigator# 48962, České Budějovice
  - Site Reference ID/Investigator# 44939, Ostrava
  - Site Reference ID/Investigator# 44936, Prague
  - Site Reference ID/Investigator# 44938, Uherské Hradiště
  - Site Reference ID/Investigator# 48963, Zlín
- Germany (5):
  - Site Reference ID/Investigator# 44941, Berlin
  - Site Reference ID/Investigator# 44945, Buch
  - Site Reference ID/Investigator# 44942, Munich
  - Site Reference ID/Investigator# 44944, Ratingen
  - Site Reference ID/Investigator# 44943, Zerbst
- Poland (5):
  - Site Reference ID/Investigator# 44946, Bydgoszcz
  - Site Reference ID/Investigator# 44982, Lodz
  - Site Reference ID/Investigator# 46584, Torun
  - Site Reference ID/Investigator# 44984, Warsaw
  - Site Reference ID/Investigator# 44983, Warsaw
- Puerto Rico (5):
  - Site Reference ID/Investigator# 38975, Caguas
  - Site Reference ID/Investigator# 40122, San Juan
  - Site Reference ID/Investigator# 39693, San Juan
  - Site Reference ID/Investigator# 38916, San Juan
  - Site Reference ID/Investigator# 39692, Vega Baja
- Spain (4):
  - Site Reference ID/Investigator# 44947, A Coruña
  - Site Reference ID/Investigator# 44987, Elche (Alicante)
  - Site Reference ID/Investigator# 44948, Oviedo (Asturias)
  - Site Reference ID/Investigator# 47782, Valencia

REFERENCES:
- [Derived] Goss SL, Klein CE, Jin Z, Locke CS, Rodila RC, Kupper H, Burmester GR, Awni WM. Methotrexate Dose in Patients With Early Rheumatoid Arthritis Impacts Methotrexate Polyglutamate Pharmacokinetics, Adalimumab Pharmacokinetics, and Efficacy: Pharmacokinetic and Exposure-response Analysis of the CONCERTO Trial. Clin Ther. 2018 Feb;40(2):309-319. doi: 10.1016/j.clinthera.2018.01.002. PMID 29402521
- [Derived] Burmester GR, Kaeley GS, Kavanaugh AF, Gabay C, MacCarter DK, Nash P, Takeuchi T, Goss SL, Rodila R, Chen K, Kupper H, Kalabic J. Treatment efficacy and methotrexate-related toxicity in patients with rheumatoid arthritis receiving methotrexate in combination with adalimumab. RMD Open. 2017 Sep 17;3(2):e000465. doi: 10.1136/rmdopen-2017-000465. eCollection 2017. PMID 28955494
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Started | 98 | 100 | 99 | 98
Completed | 83 | 93 | 93 | 89
Not Completed | 15 | 7 | 6 | 9
Not completed — Adverse Event | 3 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 7 | 5 | 2 | 3
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1
Not completed — Other Reason | 3 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX | Total
Number analyzed (Participants) | 98 | 100 | 99 | 98 | 395
Age Continuous [Mean (Standard Deviation); unit: years] | 52.0 (13.19) | 49.7 (13.14) | 52.1 (12.94) | 53.8 (14.41) | 51.9 (13.46)
Age, Customized [Number; unit: participants]
  < 65 years | 84 | 89 | 85 | 77 | 335
  > 65 years | 14 | 11 | 14 | 21 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 78 | 78 | 74 | 300
  Male | 28 | 22 | 21 | 24 | 95
28-Joint Disease Activity Score of C-reactive Protein (DAS28[CRP]) [Mean (Standard Deviation); unit: scores on a scale] — The DAS28(CRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. Baseline values are presented for 96, 98, 95, 97 participants in the 2.5 mg, 5 mg, 10 mg, and 20 mg treatment groups, respectively.
  scores on a scale | 6.10 (0.921) | 6.22 (0.943) | 5.86 (0.971) | 5.91 (1.014) | 6.02 (0.970)
Modified Total Sharp Score (mTSS) [Mean (Standard Deviation); unit: score] — MTSS is a measure of change in joint health from digitized images of radiographs of hands and feet. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). Baseline values are presented for 96, 98, 98, 95 participants in the 2.5 mg, 5 mg, 10 mg, and 20 mg treatment groups, respectively.
  score | 9.79 (12.849) | 8.60 (8.912) | 10.76 (13.017) | 10.55 (12.852) | 9.92 (12.005)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — HAQ-DI consists of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week as: without any difficulty (0); with some difficulty (1); with much difficulty (2); unable to do (3). Scores on each task were summed and averaged to provide an overall score from 0 to 3, where 0=no disability and 3=very severe, high-dependency disability. Baseline values are presented for 96, 98, 97, 98 participants in the 2.5 mg, 5 mg, 10 mg, and 20 mg treatment groups, respectively.
  units on a scale | 1.49 (0.737) | 1.57 (0.624) | 1.62 (0.667) | 1.58 (0.653) | 1.57 (0.670)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 28-Joint Disease Activity Score of C-reactive Protein (DAS28[CRP]) Low Disease Activity at Week 26
Description: Percentage of participants achieving low disease activity as defined by a clinical response (DAS28[CRP] < 3.2). The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 42.9 | 44.0 | 56.6 | 60.2

2. Secondary Outcome: Percentage of Participants With DAS28(CRP) Remission at Week 26
Description: Disease remission was defined as a disease activity score, based on CRP, for 28 joints that was < 2.6 (DAS28[CRP] < 2.6). The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10.
Time Frame: Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 27.6 | 32.0 | 37.4 | 44.9

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Criteria Response at Week 26
Description: Response, as defined by ACR 20 criteria at Week 26. A participant is a responder if the following 3 criteria for improvement from Baseline are met: ≥ 20% improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Disability Index of the Health Assessment Questionnaire
  * Acute phase reactant value (C-reactive protein).
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 67.3 | 74.0 | 76.8 | 79.6

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50 Criteria Response at Week 26
Description: Response, as defined by ACR 50 criteria at Week 26. A participant is a responder if the following 3 criteria for improvement from Baseline are met: ≥ 50% improvement in tender joint count; ≥ 50% improvement in swollen joint count; and ≥ 50% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Disability Index of the Health Assessment Questionnaire
  * Acute phase reactant value (C-reactive protein).
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 45.9 | 51.0 | 53.5 | 62.2

5. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70 Criteria Response at Week 26
Description: Response, as defined by ACR 70 criteria at Week 26. A participant is a responder if the following 3 criteria for improvement from Baseline are met: ≥ 70% improvement in tender joint count; ≥ 70% improvement in swollen joint count; and ≥ 70% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Disability Index of the Health Assessment Questionnaire
  * Acute phase reactant value (C-reactive protein).
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 24.5 | 34.0 | 41.4 | 45.9

6. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 90 Criteria Response at Week 26
Description: Response, as defined by ACR 90 criteria at Week 26. A participant is a responder if the following 3 criteria for improvement from Baseline are met: ≥ 90% improvement in tender joint count; ≥ 90% improvement in swollen joint count; and ≥ 90% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Disability Index of the Health Assessment Questionnaire
  * Acute phase reactant value (C-reactive protein).
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 7.1 | 10.0 | 17.2 | 16.3

7. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 100 Criteria Response at Week 26
Description: Response, as defined by ACR 100 criteria at Week 26. A participant is a responder if the following 3 criteria for improvement from Baseline are met: ≥ 100% improvement in tender joint count; ≥ 100% improvement in swollen joint count; and ≥ 100% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Disability Index of the Health Assessment Questionnaire
  * Acute phase reactant value (C-reactive protein).
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 1.0 | 1.0 | 2.0 | 4.1

8. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 26
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability. HAQ remission indicating normal physical function is defined by HAQ-DI score of < 0.5. Negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population with non-missing baseline and at least 1 non-missing post-baseline value (baseline is defined as the last non-missing value prior to the first dose of study drug); last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 96 | 98 | 96 | 98
units on a scale | -0.72 (0.664) | -0.71 (0.717) | -0.78 (0.647) | -0.82 (0.698)

9. Secondary Outcome: Percentage of Participants With a Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) ≤ -0.22 at Week 26
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is a change from Baseline of ≥ 0.22. HAQ remission indicating normal physical function is defined by HAQ-DI score of < 0.5. Negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 68.4 | 70.0 | 73.7 | 77.6

10. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 26
Description: The modified Total Sharp Score (mTSS) is a measure of change in joint health from digitized images of radiographs of hands and feet. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population with available data at time point (observed cases).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 88 | 94 | 95 | 90
score on a scale | 0.9 (5.62) | 0.3 (1.92) | 0.4 (3.17) | 0.2 (2.22)

11. Secondary Outcome: Percentage of Participants With No Radiographic Progression at Week 26
Description: "No radiographic progression" was defined as a change from Baseline in modified Total Sharp Score (mTSS) at Week 26 of ≤ 0.5. mTSS is a measure of change in joint health from digitized images of radiographs of hands and feet. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline, Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 64.3 | 72.0 | 76.8 | 77.6

12. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Remission at Week 26
Description: SDAI is a measure of disease activity derived as follows: SDAI = SJC28 + TJC28 + GH (cm) + PhGA (cm) + CRP (mg/dL), where TJC28 and SJC28 represent total tender joint count and total swollen joint count, respectively, based on 28 joints (including the left and right side of the body), GH = Patient's Global Assessment of Disease Activity, and PhGA = Physician's Global Assessment of Disease Activity (both measured on a visual analogue scale with a range of 0 [none] to 10 [severe]), and CRP is C-reactive protein measured in mg/dL. SDAI total score = 0 to 86. SDAI ≤ 3.3 indicates disease remission, > 3.4 to 11 = low disease activity, > 11 to 26 = moderate disease activity, and > 26 = high disease activity.
Time Frame: Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 11.2 | 22.0 | 28.3 | 29.6

13. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Remission at Week 26
Description: CDAI is a measure of disease activity derived as follows: CDAI = SJC28 + TJC28 + GH (cm) + PhGA (cm) where TJC28 and SJC28 represent total tender joint count and total swollen joint count, respectively, based on 28 joints (including the left and right side of the body), GH = Patient's Global Assessment of Disease Activity, and PhGA = Physician's Global Assessment of Disease Activity (both measured on a visual analogue scale with a range of 0 [none] to 10 [severe]). CDAI total score = 0 to 76. CDAI ≤ 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity, and > 22 = high disease activity.
Time Frame: Week 26
Population: Intent-to-Treat population; participants with a missing response were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Number analyzed (Participants) | 98 | 100 | 99 | 98
percentage of participants | 12.2 | 22.0 | 29.3 | 27.6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events and serious adverse events, defined as those that began after the first dose of study drug, but within 70 days after the last dose of study drug. Duration of treatment was 24 weeks for ADA and 25 weeks for MTX.
Arm/Group | ADA + 2.5 mg MTX | ADA + 5 mg MTX | ADA + 10 mg MTX | ADA + 20 mg MTX
Serious Adverse Events (participants affected / at risk) | 5/98 | 2/100 | 3/99 | 7/98
Other Adverse Events (participants affected / at risk) | 24/98 | 26/100 | 34/99 | 41/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADA + 2.5 mg MTX (N=98) | ADA + 5 mg MTX (N=100) | ADA + 10 mg MTX (N=99) | ADA + 20 mg MTX (N=98)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ASTHENIA (General disorders) | 1 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADA + 2.5 mg MTX (N=98) | ADA + 5 mg MTX (N=100) | ADA + 10 mg MTX (N=99) | ADA + 20 mg MTX (N=98)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 5 | 4 | 4
DIARRHOEA (Gastrointestinal disorders) | 3 | 6 | 6 | 3
NAUSEA (Gastrointestinal disorders) | 7 | 5 | 13 | 8
FATIGUE (General disorders) | 2 | 2 | 6 | 4
NASOPHARYNGITIS (Infections and infestations) | 3 | 6 | 6 | 11
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 2 | 3 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 0
DIZZINESS (Nervous system disorders) | 4 | 0 | 6 | 4
HEADACHE (Nervous system disorders) | 4 | 6 | 5 | 9
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 5 | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.